CLINICAL TRIAL: NCT06363656
Title: Assessment of Smartwatch SAMSUNG to Monitor Sleep Quality: an Observational Prospective Study - SleepEx2 Protocol
Acronym: SLEEP-EX2
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Geraldo Lorenzi Filho, Director, Head of the Sleep Laboratory, Principal Investigator, Associate Professor, University of Sao Paulo General Hospital
Other Study IDs: 76455623.5.0000.0068
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Insomnia; Sleep Initiation and Maintenance Disorders; Health Status; Wearable Electronic Devices; Sleep
Keywords: Wearable Electronic Devices; Insomnia; Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- single-group: Participants who declare having problems with sleeping/insomnia
  Interventions: Device: Wears the smartwatch during the sleep time to capture sleep characteristics and answer questionaires

INTERVENTIONS:
Device: Wears the smartwatch during the sleep time to capture sleep characteristics and answer questionaires — * Synchronization of smartwatch with smartphone (internet connection) to send sleep characteristics captured by the application
  * Weight
  * Height
  * Body measurements (circumferences)
  * Questionnaires about overall health status
  * Pittsburgh Sleep Quality Index questionnaire
  * Insomnia Severity Index
  * Sleep Hygiene Index
  * Epworth Sleepiness Scale
  * NoSAS score (Neck, Obesity, Snoring, Age, Sex)

SUMMARY:
The goal of this study is to learn if a smartwatch is effective to identify factors related to sleep quality and habits of adults (30 years old or more), enabling the improvement and/or creation of instruments to assess overall health status and sleep quality.

The main question it aims to answer is:

- Does the smartwatch application (software) indicate sleep habits and measure sleep quality in accordance to the standardized clinical instruments commonly used to assess sleep?

DETAILED DESCRIPTION:
Participants will answer questionnaires about overall health status, sleep quality and insomnia at the beginning, at 16 days follow-up, and at the end of the study. Participants must use the smartwatch for at least a 12-hour period that includes night time, during a minimum of 30 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Adults (30 years old or more);
* Minimum score of 7 on Pittsburgh Sleep Quality Index;
* Capable of giving consent.

Exclusion Criteria:

* Night shift workers;
* Skin condition that may interfere with optic sensor readings - such as Lupus, Atopic Dermatitis, Vitiligo;
* Tattoo on the wrist area that may interfere with optic sensor readings;
* Allergies or sensitivities to the components/materials of the smartwatch;
* Health condition that may be considered risky/unsafe by the medical team;
* Pregnant women.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any participant that reports sleep problems or insomnia screened by the open survey sent to different groups in the city of Sao Paulo (Brazil).
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Concordance between the smartwatch application and clinical assessment | 1) at the beginning (start); 2) at the 16-days follow-up (middle); 3) at the 30-days follow-up (end).
  Intraclass correlation coefficient calculated between sleep characteristics captured by the smartwatch and scores of all questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Geraldo Lorenzi Filho, MD, PhD, Principal Investigator — Sleep Laboratory, Instituto do Coração, Hospital das Clínicas HCFMUSP
Locations (1):
- Instituto do Coracao do Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Massoomi MR, Handberg EM. Increasing and Evolving Role of Smart Devices in Modern Medicine. Eur Cardiol. 2019 Dec 18;14(3):181-186. doi: 10.15420/ecr.2019.02. eCollection 2019 Dec. PMID 31933689
- [Background] Knutson KL, Phelan J, Paskow MJ, Roach A, Whiton K, Langer G, Hillygus DS, Mokrzycki M, Broughton WA, Chokroverty S, Lichstein KL, Weaver TE, Hirshkowitz M. The National Sleep Foundation's Sleep Health Index. Sleep Health. 2017 Aug;3(4):234-240. doi: 10.1016/j.sleh.2017.05.011. Epub 2017 Jun 20. PMID 28709508
- [Background] Kasai T, Floras JS, Bradley TD. Sleep apnea and cardiovascular disease: a bidirectional relationship. Circulation. 2012 Sep 18;126(12):1495-510. doi: 10.1161/CIRCULATIONAHA.111.070813. No abstract available. PMID 22988046
- [Background] Allen J. Photoplethysmography and its application in clinical physiological measurement. Physiol Meas. 2007 Mar;28(3):R1-39. doi: 10.1088/0967-3334/28/3/R01. Epub 2007 Feb 20. PMID 17322588
- [Background] Perez MV, Mahaffey KW, Hedlin H, Rumsfeld JS, Garcia A, Ferris T, Balasubramanian V, Russo AM, Rajmane A, Cheung L, Hung G, Lee J, Kowey P, Talati N, Nag D, Gummidipundi SE, Beatty A, Hills MT, Desai S, Granger CB, Desai M, Turakhia MP; Apple Heart Study Investigators. Large-Scale Assessment of a Smartwatch to Identify Atrial Fibrillation. N Engl J Med. 2019 Nov 14;381(20):1909-1917. doi: 10.1056/NEJMoa1901183. PMID 31722151
- [Background] Fonseca P, Weysen T, Goelema MS, Most EIS, Radha M, Lunsingh Scheurleer C, van den Heuvel L, Aarts RM. Validation of Photoplethysmography-Based Sleep Staging Compared With Polysomnography in Healthy Middle-Aged Adults. Sleep. 2017 Jul 1;40(7). doi: 10.1093/sleep/zsx097. PMID 28838130
- [Background] Bertolazi AN, Fagondes SC, Hoff LS, Dartora EG, Miozzo IC, de Barba ME, Barreto SS. Validation of the Brazilian Portuguese version of the Pittsburgh Sleep Quality Index. Sleep Med. 2011 Jan;12(1):70-5. doi: 10.1016/j.sleep.2010.04.020. Epub 2010 Dec 9. PMID 21145786
- [Background] Tonon AC, Amando GR, Carissimi A, Freitas JJ, Xavier NB, Caumo GH, Silva LG, de Souza DOG, Hidalgo MP. The Brazilian-Portuguese version of the Sleep Hygiene Index (SHI): validity, reliability and association with depressive symptoms and sleep-related outcomes. Sleep Sci. 2020 Jan-Mar;13(1):37-48. doi: 10.5935/1984-0063.20190130. PMID 32670491
- [Background] Bertolazi AN, Fagondes SC, Hoff LS, Pedro VD, Menna Barreto SS, Johns MW. Portuguese-language version of the Epworth sleepiness scale: validation for use in Brazil. J Bras Pneumol. 2009 Sep;35(9):877-83. doi: 10.1590/s1806-37132009000900009. English, Portuguese. PMID 19820814
- [Background] Castro LS. Adaptação e validação do Índice de Gravidade de Insônia (IGI): Caracterização Populacional, Valores Normativos e Aspectos Associados 2011 [Available from: http://repositorio.unifesp.br/handle/11600/23193.
- [Background] Coutinho Costa J, Rebelo-Marques A, Machado JN, Gama JMR, Santos C, Teixeira F, Moita J. Validation of NoSAS (Neck, Obesity, Snoring, Age, Sex) score as a screening tool for obstructive sleep apnea: Analysis in a sleep clinic. Pulmonology. 2019 Sep-Oct;25(5):263-270. doi: 10.1016/j.pulmoe.2019.04.004. Epub 2019 Jun 10. PMID 31196834
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660